CLINICAL TRIAL: NCT00159757
Title: 12 Week Open Label, Multicenter, Non-Comparative Switch Study Evaluating Efficacy, Tolerability And Safety Of Oral Ziprasidone In Treatment Of Patients Suffering From Schizophrenia Who Have Already Been Treated With An Other Antipsychotic.
Brief Title: 12 Week Open, Non-Comparative Switch Study Of Oral Ziprazidone In Previously Treated Schizophrenic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description for Termination Reason
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281122
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone

INTERVENTIONS:
Drug: ziprazidone

SUMMARY:
There has been evidence that ziprasidone is efficacious in decreasing the magnitude of both positive and negative symptoms of schizophrenia, and also effective in the treatment of depressive symptoms. It shows good tolerance with low incidence of extrapyramidal side effects and does not significantly influence body weight. As it has been shown that ziprasidone is efficacious and safe in patients who have been pretreated with other antipsychotic that has to be withdrawn either due to the side effects or not satisfied efficacy. The purpose of the study was to provide further evidence for the efficacy and safety of patients with schizophrenia and allow for psychiatrists in Hungary to gain experience with the drug before wide commercial availability.

DETAILED DESCRIPTION:
Study was terminated due to difficulty in enrolling the targeted number of patients on March 1, 2005, last subject last visit date was Feb.16, 2005. There were no safety concerns involved in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of schizophrenia according to DSM-IV-IV from patient's medical files
* subjects with current treatment with typical or atypical neuroleptics which should be changed

Exclusion Criteria:

* patients with significant cardiovascular illness (recent acute myocardial infarction, uncompensated heart failure, cardiac arrhythmia)
* in the patients' history clinically significant ECG abnormalities particularly prolongation of QT interval of more than 500 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-11; Study Completion 2005-02

PRIMARY OUTCOMES:
Efficacy- To assess the syndromes of the psychosis expressed as the PANSS total score
Safety- Incidence and severity of the side effects

SECONDARY OUTCOMES:
To assess the change of the clinical impression in CGI (Clinical Global Impression of Change scale)
To evaluate the influence on the body weight change.
To assess the subject's view on the treatment with ziprasidone
To assess the subject's antidepressive efficacy by Calgary and Hamilton depression scales

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Hungary (8):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Esztergom
  - Pfizer Investigational Site, Kecskemét
  - Pfizer Investigational Site, Kistarcsa
  - Pfizer Investigational Site, Pécs
  - Pfizer Investigational Site, Székesfehérvár
  - Pfizer Investigational Site, Tatabánya

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281122&StudyName=12+Week+Open%2C+Non%2DComparative+Switch+Study+Of+Oral+Ziprazidone+In+Previously+Treated+Schizophrenic+Patients